CLINICAL TRIAL: NCT00970268
Title: A Long-term, Randomized, Double-blind Extension Study of the Safety, Tolerability, and Efficacy of Aclidinium Bromide at Two Dose Levels When Administered to Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease
Brief Title: Long-term Extension Study of the Safety, Tolerability, and Efficacy of Aclidinium Bromide in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD) (LAS-MD-36)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LAS-MD-36
Record Dates: First submitted 2009-09-01; First posted 2009-09-02 (Estimated); Results first posted 2012-09-14 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Chronic Obstructive Pulmonary Disease; Chronic Bronchitis; Emphysema; Airflow Obstruction, Chronic; Chronic Airflow Obstruction; Chronic Obstructive Airway Disease; Chronic Obstructive Lung Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic; Emphysema | interventions — aclidinium bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Aclidinium bromide dose, inhaled, for 52 weeks of treatment
  Interventions: Drug: Aclidinium bromide
- 2 (Experimental): Aclidinium bromide dose, inhaled, for 52 weeks of treatment
  Interventions: Drug: Aclidinium bromide

INTERVENTIONS:
Drug: Aclidinium bromide — Aclidinium bromide 200 μg, oral inhalation twice per day for 52 weeks of treatment
  Arms: 1
Drug: Aclidinium bromide — Aclidinium bromide 400 μg, oral inhalation twice per day for 52 weeks of treatment
  Arms: 2

SUMMARY:
The purpose of this extension study is to evaluate the long-term safety, tolerability, and efficacy of inhaled aclidinium bromide at two dose levels in patients with moderate to severe chronic obstructive pulmonary disease (COPD). This study will be 54 weeks in duration; a 52-week double-blind treatment period and 2 week follow-up phone call, following a 12 week lead-in study. All patients will be randomized from the lead-in study at one of two doses of aclidinium.

ELIGIBILITY:
Inclusion Criteria:

* Completion of a lead-in study (NCT00891462)

Exclusion Criteria:

* Use or anticipated use of any medication prohibited in this study
* Evidence of abnormal clinical laboratory values, vital signs, or electrocardiographic (ECG) results or the presence of abnormities in physical examination findings
* The presence of anti-cholinergic effects (eg, dry mouth, urinary retention, narrow angle glaucoma)
* QTcB of >500 msec on both the pre-dose and post-dose ECG
* Women who are pregnant, intend to become pregnant, or are breast-feeding
* A life expectancy of less than 1 year
* Noncompliance with IP dosing and/or attending clinic visits during the lead-in study
* Significant interruption of double-blind therapy during the transition from the lead-in study into the extension study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2009-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esther Garcia, MD, Study Director — AstraZeneca
Locations (83):
- United States (77):
  - Forest Investigative Site 1162, Birmingham, Alabama
  - Forest Investigative Site 1127, Mobile, Alabama
  - Forest Investigative Site 0909, Glendale, Arizona
  - Forest Investigative Site 2060, Phoenix, Arizona
  - Forest Investigative Site 2065, Fullerton, California
  - Forest Investigative Site 1088, Lakewood, California
  - Forest Investigative Site 1122, Orange, California
  - Forest Investigative Site 2029, Rancho Mirage, California
  - Forets Investigative Site 2064, Riverside, California
  - Forest Investigative Site 0517, Sacramento, California
  - Forest Investigative Site 2009, San Diego, California
  - Forest Investigative Site 1137, Colorado Springs, Colorado
  - Forest Investigative Site 2100, Waterbury, Connecticut
  - Forest Investigative Site 1154, Brandon, Florida
  - Forest Investigative Site 1152, Clearwater, Florida
  - Forest Investigative Site 0670, DeLand, Florida
  - Forest Investigative Site 0990, Fort Lauderdale, Florida
  - Forest Investigative Site 1167, Melbourne, Florida
  - Forest Investigative Site 1060, Ormond Beach, Florida
  - Forest Investigative Site 0974, Pensacola, Florida
  - Forest Investigative Site 2082, Tamarac, Florida
  - Forest Investigative Site 2053, Tampa, Florida
  - Forest Investigative Site 2047, Tampa, Florida
  - Forest Investigative Site 1185, Winter Park, Florida
  - Forest Investigative Site 1183, Atlanta, Georgia
  - Forest Investigative Site 0987, Austell, Georgia
  - Forest Investigative Site 1101, Blue Ridge, Georgia
  - Forest Investigative Site 1180, Decatur, Georgia
  - Forest Investigative Site 1161, Duluth, Georgia
  - Forest Investigative Site 2051, River Forest, Illinois
  - Forest Investigative Site 0989, Skokie, Illinois
  - Forest Investigative Site 1149, South Bend, Indiana
  - Forest Investigative Site 2085, Crescent Springs, Kentucky
  - Forest Investigative Site 0539, Lexington, Kentucky
  - Forest Investigative Site 2024, Lafayette, Louisiana
  - Forest Investigative Site 2040, Biddeford, Maine
  - Forest Investigative Site 1128, Edina, Minnesota
  - Forest Investigative Site 2041, Minneapolis, Minnesota
  - Forest Investigative Site 1124, Minneapolis, Minnesota
  - Forest Investigative Site 1100, Florissant, Missouri
  - Forest Investigative Site 2079, Saint Charles, Missouri
  - Forest Investigative Site 2067, Butte, Montana
  - Forest Investigative Site 1169, Papillion, Nebraska
  - Forest Investigative Site 1150, Berlin, New Jersey
  - Forest Investigative Site 2084, Summit, New Jersey
  - Forest Investigative Site 1147, Brooklyn, New York
  - Forest Investigative Site 1119, Elmira, New York
  - Forest Investigative Site 1151, New Hyde Park, New York
  - Forest Investigative Site 1141, New York, New York
  - Forest Investigative Site 1163, New York, New York
  - Forest Investigative Site 1130, Asheville, North Carolina
  - Forest Investigative Site 1134, Canton, Ohio
  - Forest Investigative Site 1181, Centerville, Ohio
  - Forest Investigative Site 1136, Cincinnati, Ohio
  - Forest Investigative Site 2007, Cincinnati, Ohio
  - Forest Investigative Site 2028, Cincinnati, Ohio
  - Forest Investigative Site 0959, Columbus, Ohio
  - Forest Investigative Site 2006, Columbus, Ohio
  - Forest Investigative Site 2043, Medford, Oregon
  - Forest Investigative Site 1106, Portland, Oregon
  - Forest Investigative Site 1126, Bethlehem, Pennsylvania
  - Forest Investigative Site 2016, Erie, Pennsylvania
  - Forest Investigative Site 1146, Pittsburgh, Pennsylvania
  - Forest Investigative Site 1158, Upland, Pennsylvania
  - Forest Investigative Site 1089, East Providence, Rhode Island
  - Forest Investigative Site 1144, Johnston, Rhode Island
  - Forest Investigative Site 2072, Charleston, South Carolina
  - Forest Investigative Site 1078, Greenville, South Carolina
  - Forest Investigative Site 2080, Greer, South Carolina
  - Forest Investigative Site 1121, Spartanburg, South Carolina
  - Forest Investigative Site 1155, Dallas, Texas
  - Forest Investigative Site 2012, Fort Worth, Texas
  - Forest Investigative Site 1165, San Antonio, Texas
  - Forest Investigative Site 1129, Waco, Texas
  - Forest Investigative Site 2099, Richmond, Virginia
  - Forest Investigative Site 1142, Spokane, Washington
  - Forest Investigative Site 0988, Tacoma, Washington
- Canada (6):
  - Forest Investigative Site 2201, Kelowna, British Columbia
  - Forest Investigative Site 1177, Vancouver, British Columbia
  - Forest Investigative Site 2200, Niagara Falls, Ontario
  - Forest Investigative Site 1168, Toronto, Ontario
  - Forest Investigative Site 1171, Toronto, Ontario
  - Forest Investigative Site 2203, Toronto, Ontario

REFERENCES:
- [Derived] D'Urzo A, Kerwin E, Rennard S, He T, Gil EG, Caracta C. One-year extension study of ACCORD COPD I: safety and efficacy of two doses of twice-daily aclidinium bromide in patients with COPD. COPD. 2013 Aug;10(4):500-10. doi: 10.3109/15412555.2013.791809. Epub 2013 May 16. PMID 23679347

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient recruitment occurred from August of 2009 to March of 2010 and was by invitation only to patients who had completed study NCT00891462 (LAS-MD-33). In total, there were 77 individual study sites, 71 in the United States and 6 additional sites in Canada.
Pre-assignment Details: From the total of 291 patients enrolled, 289 patients (99.3%) received at least 1 dose of double-blind treatment and therefore were included in the Safety Population. Of these patients, 246 (84.5%) had a baseline and at least 1 postbaseline FEV1 assessment and qualified for the Intent To Treat (ITT) Population.
Groups:
- Aclidinium Bromide 200 μg: Aclidinium bromide, 200 microgram dose, oral inhalation twice per day for 52 weeks of treatment.
- Aclidinium Bromide 400 μg: Aclidinium bromide, 400 microgram dose, oral inhalation twice per day for 52 weeks of treatment.
Period: Overall Study
Arm/Group | Aclidinium Bromide 200 μg | Aclidinium Bromide 400 μg
Started | 139 | 152
Completed | 96 | 103
Not Completed | 43 | 49
Not completed — Withdrawal by Subject | 12 | 19
Not completed — Adverse Event | 15 | 12
Not completed — Lack of Efficacy | 3 | 6
Not completed — Protocol Violation | 4 | 7
Not completed — Other Reason | 3 | 1
Not completed — COPD Exacerbation | 4 | 2
Not completed — Lost to Follow-up | 1 | 2
Not completed — Inclusion/Exclusion Criteria | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aclidinium Bromide 200 μg | Aclidinium Bromide 400 μg | Total
Number analyzed (Participants) | 137 | 152 | 289
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (10.1) | 64.4 (10.0) | 63.9 (9.9)
Age, Customized [Number; unit: participants]
  ≥ 40 to < 60 years | 49 | 40 | 89
  ≥ 60 to < 70 years | 51 | 67 | 118
  ≥ 70 years | 37 | 45 | 82
Gender [Count of Participants; unit: Participants]
  Female | 63 | 76 | 139
  Male | 74 | 76 | 150
Region of Enrollment [Number; unit: participants]
  United States | 128 | 138 | 266
  Canada | 9 | 14 | 23

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Morning Pre-dose (Trough) Forced Expiratory Volume in One Second (FEV1)
Description: Change From Baseline (Visit 2 of lead-in Study NCT00891462, [LAS-MD-33]) to Week 52 (Week 64 From Start of NCT00891462, [LAS-MD-33]) in Morning Predose (Trough) FEV1
Time Frame: Change from baseline (visit 2 of lead-in study LAS-MD-33) to 52 weeks
Population: From the total of 291 patients enrolled, 289 patients (99.3%) received at least 1 dose of double-blind treatment and therefore were included in the Safety Population. Of these patients, 246 (84.5%) had a baseline and at least 1 postbaseline FEV1 assessment and qualified for the ITT Population
Measure: Least Squares Mean (Standard Error); unit: L
Groups:
- Placebo - Aclidinium Bromide 200 μg: Aclidinium bromide, 200 microgram dose, oral inhalation twice per day for 52 weeks of treatment for patients who received 12 weeks of placebo in the lead-in study.
- Aclidinium Bromide 200 μg - Aclidinium Bromide 200 μg: Aclidinium bromide, 200 microgram dose, oral inhalation twice per day for 52 weeks of treatment in patients who also received 200 micrograms of Aclidinium bromide for 12 weeks in the lead-in study.
- Placebo - Aclidinium Bromide 400 μg: Aclidinium bromide, 400 microgram dose, oral inhalation, twice per day for 52 weeks of treatment for patients who received 12 weeks of placebo in the lead-in study.
- Aclidinium Bromide 400 μg - Aclidinium Bromide 400 μg: Aclidinium bromide, 400 microgram dose, oral inhalation twice per day for 52 weeks of treatment in patients who also received 400 microgram of Aclidinium bromide for 12 weeks in the lead-in study.
Arm/Group | Placebo - Aclidinium Bromide 200 μg | Aclidinium Bromide 200 μg - Aclidinium Bromide 200 μg | Placebo - Aclidinium Bromide 400 μg | Aclidinium Bromide 400 μg - Aclidinium Bromide 400 μg
Number analyzed (Participants) | 38 | 76 | 41 | 91
L | -0.035 (0.040) | 0.069 (0.028) | 0.069 (0.037) | 0.056 (0.025)

2. Secondary Outcome: Change From Baseline in Peak FEV1
Description: Change From Baseline (Visit 2 of study NCT00891462, [LAS-MD-33])in Peak FEV1 in liters at Week 52 (Week 64 from the start of NCT00891462, [LAS-MD-33]).
Time Frame: 52 weeks
Measure: Least Squares Mean (Standard Error); unit: L
Groups:
- Placebo - Aclidinium Bromide 400 μg: Aclidinium bromide, 400 microgram dose, oral inhalation twice per day for 52 weeks of treatment for patients who received 12 weeks of placebo in the lead-in study.
- Aclidinium Bromide 400 μg - Aclidinium Bromide 400 μg: Aclidinium bromide, 400 microgram dose, oral inhalation twice per day for 52 weeks of treatment in patients who also received 400 micrograms of Aclidinium bromide for 12 weeks in the lead-in study.
Arm/Group | Placebo - Aclidinium Bromide 200 μg | Aclidinium Bromide 200 μg - Aclidinium Bromide 200 μg | Placebo - Aclidinium Bromide 400 μg | Aclidinium Bromide 400 μg - Aclidinium Bromide 400 μg
Number analyzed (Participants) | 38 | 76 | 41 | 91
L | 0.111 (0.040) | 0.213 (0.028) | 0.222 (0.038) | 0.219 (0.025)

ADVERSE EVENTS:
Time Frame: Adverse Event Reporting occurred from August 2009 to November 2010 at 77 study sites (71 in the United States and 6 additional sites in Canada).
Groups:
- Placebo to Aclidinium Bromide 200 μg: Patients were given 12 weeks of placebo, then switched to Aclidinium bromide, 200 microgram dose, oral inhalation twice per day for 52 weeks of treatment
- Aclidinium Bromide 200 μg to Aclidinium Bromide 200 μg: Patients were given 12 weeks of Aclidinium bromide, 200 microgram dose, then continued with the 200 microgram dose, oral inhalation twice per day for an additional 52 weeks of treatment.
- Placebo to Aclidinium Bromide 400μg: Patients were given 12 weeks of placebo, then switched to Aclidinium bromide, 400 microgram dose, oral inhalation twice per day for 52 weeks of treatment
- Aclidinium Bromide 400μg to Aclidinium Bromide 400μg: Patients were given 12 weeks of Aclidinium bromide, 400 microgram dose, then continued with the 400 microgram dose twice per day, oral inhalation, for an additional 52 weeks of treatment.
Arm/Group | Placebo to Aclidinium Bromide 200 μg | Aclidinium Bromide 200 μg to Aclidinium Bromide 200 μg | Placebo to Aclidinium Bromide 400μg | Aclidinium Bromide 400μg to Aclidinium Bromide 400μg
Serious Adverse Events (participants affected / at risk) | 7/44 | 13/93 | 7/46 | 13/106
Other Adverse Events (participants affected / at risk) | 36/44 | 63/93 | 28/46 | 64/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo to Aclidinium Bromide 200 μg (N=44) | Aclidinium Bromide 200 μg to Aclidinium Bromide 200 μg (N=93) | Placebo to Aclidinium Bromide 400μg (N=46) | Aclidinium Bromide 400μg to Aclidinium Bromide 400μg (N=106)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1 | 6
Pneumonia (Infections and infestations) | 1 | 3 | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Dyspepsia (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Multiple drug overdose accidental (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo to Aclidinium Bromide 200 μg (N=44) | Aclidinium Bromide 200 μg to Aclidinium Bromide 200 μg (N=93) | Placebo to Aclidinium Bromide 400μg (N=46) | Aclidinium Bromide 400μg to Aclidinium Bromide 400μg (N=106)
Chronic obstructive pulmonary disorder (Respiratory, thoracic and mediastinal disorders) | 16 | 23 | 14 | 24
Bundle branch block left (Cardiac disorders) | 3 | 3 | 0 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 0 | 1 | 2
Nausea (Gastrointestinal disorders) | 4 | 1 | 1 | 2
Fatigue (General disorders) | 4 | 3 | 0 | 3
Pyrexia (General disorders) | 3 | 0 | 0 | 3
Nasopharyngitis (Infections and infestations) | 4 | 8 | 4 | 10
Urinary tract infection (Infections and infestations) | 4 | 4 | 3 | 8
Upper respiratory tract infection (Infections and infestations) | 5 | 6 | 2 | 6
Bronchitis (Infections and infestations) | 3 | 1 | 1 | 4
Sinusitis (Infections and infestations) | 5 | 6 | 1 | 3
Pneumonia (Infections and infestations) | 3 | 4 | 1 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 6 | 3 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 6 | 5 | 1
Blood glucose increased (Investigations) | 3 | 3 | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 7 | 0 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 5 | 3 | 4
Insomnia (Psychiatric disorders) | 2 | 2 | 2 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 7 | 4 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 7 | 4 | 4
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 6
Hypertension (Vascular disorders) | 3 | 4 | 1 | 3
Headache (Nervous system disorders) | 3 | 5 | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study will be the property of Forest Research Institute, Inc. An integrated clinical and statistical report will be prepared at the completion of the study.

Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and Forest Research Institute, Inc.